CLINICAL TRIAL: NCT07271329
Title: Risk-stratification of Emergency Department Suspected Sepsis (REDS) Score Versus Quick Sequential Organ Failure Assessment (qSOFA) Score to Predict Mortality in Patients With Suspected Sepsis
Brief Title: REDS SCORE VERSUS qSOFA SCORE to Predict Mortality in Patients With Suspected Sepsis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MN MohamedHussin, Resident at Emergency Department, Assiut University
Other Study IDs: Reds score versus qSOFA score
Record Dates: First submitted 2025-11-28; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Sepsis in ED Patients
MeSH Terms: interventions — Sphygmomanometers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients will be randomly assigned to two groups: 1) Group A 2)Group B: Patients will be randomly assigned to two groups:
  1. Group A: Initial vital signs upon arrival at ED triage to evaluate the REDS score [ Time Frame: Timepoint 0 (ED triage) Age: ≥ 65 years old (1 point) Altered Mental State: (1 point) [from 1-15] Respiratory Rate: ≥22 breaths/min (1point ) [yes or not] Systolic Blood Pressure: ≤100 mm Hg (1 point) [yes or not] Serum Albumin: ≤27 g/L (1 point) [yes or not] INR: ≥1.3 (1 point)[yes or not] Lactate: 2.1-3.9 mmol/L (1 point), ≥4 mmol/L (3 points) Refractory Hypotension: (2 points for lactate ≤2 mmol/L, 3 points for lactate >2 mmol/L) will be assessed to evaluate the REDS score.
  2. Group B: Initial vital signs upon arrival at ED triage to evaluate the qSOFA score [ Time Frame: Timepoint 0 (ED triage) ] .
     * Respiratory rate per minute
     * Mental status
     * Systolic blood pressure.
  Interventions: Device: Sphygmomanometer

INTERVENTIONS:
Device: Sphygmomanometer — Mercury sphygmomanometer for measuring blood pressure

SUMMARY:
Our goal in this work is to compare the predictive accuracy of the REDS score versus qSOFA in identifying in-hospital mortality among ED patients with suspected sepsis and improving outcomes in ED patients.

DETAILED DESCRIPTION:
Sepsis is a life threatening condition and a major cause of morbidity and mortality in emergency department worldwide.Patients at high-risk of death may be identified by using an evidence based risk-stratification score. The ED is a busy and hard environment and any score that is used should be easy to calculate using readily available variables. The objective criteria defining sepsis, a minimum two-point increase as in qSoFA score .

The REDS (Risk-stratification of Emergency Department suspected Sepsis) score is a tool used to assess the risk of mortality in patients with suspected sepsis in the emergency department. It combines several factors including age, altered mental state, respiratory rate, systolic blood pressure, serum albumin, INR, lactate levels, and refractory hypotension. A score of 3 or more is considered high-risk. Our goal in this work is to compare the predictive accuracy of the REDS score versus qSOFA in identifying in-hospital mortality among ED patients with suspected sepsis and improving outcomes in ED patients.

The REDS score includes the following variables, each assigned a point value:

Age: ≥ 65 years old (1 point) Altered Mental State: (1 point) Respiratory Rate: ≥ 22 breaths/min (1 point) Systolic Blood Pressure: ≤ 100 mm Hg (1 point) Serum Albumin: ≤ 27 g/L (1 point) INR: ≥ 1.3 (1 point) Lactate: 2.1-3.9 mmol/L (1 point), ≥ 4 mmol/L (3 points) Refractory Hypotension: (2 points for lactate ≤ 2 mmol/L, 3 points for lactate >2 mmol/L)

Interpreting the REDS score:

0-2: Low risk of death 3 or more: High risk of death The REDS score is a useful tool for emergency departments to quickly identify patients who may be at higher risk of mortality from sepsis and need more aggressive or immediate treatment.The quick SOFA (qSOFA) score is a bedside tool used to quickly assess the risk of death or prolonged intensive care unit stay in patients with suspected infection. It uses three criteria: respiratory rate, altered mental status, and systolic blood pressure. A score of 2 or more indicates a higher risk.

qSOFA Criteria:

1. Respiratory Rate: 22 breaths per minute or higher.
2. Altered Mental Status: A Glasgow Coma Scale score less than 15.
3. Systolic Blood Pressure: 100 mmHg or lower.

Scoring:

Each criterion met scores 1 point. A score of 2 or more indicates a higher risk of poor outcome. qSOFA helps identify patients with suspected infection who are likely to have sepsis. It is a rapid assessment tool that can be used in urgent and resource-limited settings

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 y presented to the ED with suspected or confirmed infection, both sex qSOFA criterion met on arrival ≥ 2

Exclusion Criteria:

* Patient less than 18 years Incomplete vital sign records upon ED arrival Pregnant patients Those with DNR state Immune compromised patient as leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our goal in this work is to compare the predictive accuracy of the REDS score versus qSOFA in identifying in-hospital mortality among ED patients with suspected sepsis and improving outcomes in ED patients.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | 30 day
  primary outcome will be mortality during the 30 day follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Anwar, Consultant of Anathesia ICU, Principal Investigator — Assiut University; Haitham Mohammed Ahmed, Lecturer of Anesthesia,ICU, Study Director — Assiut University
Locations (1):
- Assiut, Asyut, Abo Tig, Egypt